CLINICAL TRIAL: NCT03209076
Title: Robotic Versus Laparoscopic Low Anterior Resection for Rectal Cancer: A Randomized Study
Brief Title: Robotic Versus Laparoscopic Low Anterior Resection for Rectal Cancer
Acronym: RAR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Collaborators: Hospital de Câncer de Barretos (Other); Hospital dos Servidores do Estado do Rio de Janeiro (Other Government)
Responsible Party: Principal Investigator, Marcus Valadão, Principal Investigator, Instituto Nacional de Cancer, Brazil
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RAR Trial
Record Dates: First submitted 2017-04-10; First posted 2017-07-06 (Actual); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Rectal Neoplasms; Sexual Dysfunction; Urinary Incontinence; Quality of Life
Keywords: rectal neoplasms; sexual dysfunctions; Urinary incontinence; Quality of life; robotic surgical procedures; laparoscopy
MeSH Terms: conditions — Rectal Neoplasms; Sexual Dysfunction, Physiological; Urinary Incontinence | interventions — Robotics; Laparoscopy

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic (Experimental): Robotic low anterior resection
  Interventions: Procedure: Robotic
- Laparoscopic (Active Comparator): Laparoscopic low anterior resection
  Interventions: Procedure: Laparoscopic

INTERVENTIONS:
Procedure: Robotic — Robotic low anterior resection
  Arms: Robotic
Procedure: Laparoscopic — Laparoscopic low anterior resection
  Arms: Laparoscopic

SUMMARY:
Prospective randomized trial comparing robotic versus laparoscopic Low anterior resection for rectal cancer.

Primary endpoint: Compare urinary dysfunction between robotic and laparoscopic approach.

DETAILED DESCRIPTION:
Prospective randomized trial comparing robotic versus laparoscopic Low anterior resection for rectal cancer.

The Aim of the study is to compare two surgical approaches (robotic versus laparoscopic) for rectal cancer treatment regarding functional outcomes (sexual and urinary dysfunctions), quality of life, post operative outcomes and oncologic outcomes.

Patients with the diagnosis of T3 mid and low rectal cancer will be randomized to robotic or laparoscopic procedure after neoadjuvant chemoradiation. Quality of life questionnaires and Urodynamic test will be applied before and after the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Mid or low Rectal Adenocarcinoma
* Performance Status (ECOG) 0 - 2

Exclusion Criteria:

* Metastatic disease
* Congestive heart failure
* Renal failure
* Diabetes
* Pregnancy
* Neurologic disorders
* Alfa blockers user
* Patients who are candidates to APR ( Abdomino-perineal resection)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
Urinary dysfunction | Change from Before surgery to 3 months after surgery
  Urodynamic test

SECONDARY OUTCOMES:
Sexual dysfunction | Change from Before surgery to 3 months after surgery
  Quality of life questionnaire
Post operative outcomes | Within the first 30 days after the surgical procedure
  Post operative complications
Costs | From the surgical procedure until the last follow up, which will be 24 months or the day of death.
  Costs in Brazilian currency of each procedure

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Valadão, Dr, Principal Investigator — Instituto Nacional de Câncer-INCA
Locations (1):
- Instituto Nacional de Câncer- INCA, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Jesus JP, Valadao M, de Castro Araujo RO, Cesar D, Linhares E, Iglesias AC. The circumferential resection margins status: A comparison of robotic, laparoscopic and open total mesorectal excision for mid and low rectal cancer. Eur J Surg Oncol. 2016 Jun;42(6):808-12. doi: 10.1016/j.ejso.2016.03.002. Epub 2016 Mar 23. PMID 27038996